CLINICAL TRIAL: NCT04385602
Title: Effect of Administration of Intratracheal Dexmedetomidine on Recovery From General Anesthesia in Pediatrics Undergoing Lower Abdominal Surgery: a Randomized Double-blinded Controlled Study.
Brief Title: Effect of Intratracheal Dexmedetomidine Administration on Recovery From General Anesthesia in Pediatrics Undergoing Lower Abdominal Surgery:
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohammed AboelFadl, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: intratracheal dexmed
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Intratracheal; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Subject, Caregiver, Investigator, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CON group (Placebo Comparator): placebo
  Interventions: Drug: Saline Solution
- DT group (Active Comparator): Intratracheal dexmedetomidine
  Interventions: Drug: Intratracheal dexmedetomidine

INTERVENTIONS:
Drug: Intratracheal dexmedetomidine — Thirty minutes before the end of the surgery, Dex (0.5μg/kg diluted and mixed in 1ml saline in a medical spray bottle) will be sprayed down the intratracheal tube
  Other Names: precedex
  Arms: DT group
Drug: Saline Solution — Thirty minutes before the end of the surgery, 1ml saline in a medical spray bottle will be sprayed down the intratracheal tube
  Arms: CON group

SUMMARY:
The incidence of intratracheal tube-induced laryngeal irritation, including coughing, bucking, and cardiovascular stimulation, on emergence from general anesthesia has been reported to occur in 38% and 96% of cases. This may cause agitation and unstable hemodynamics during anesthesia recovery, and can lead to complications, such as laryngeal edema, sore throat, increased intra-abdominal pressure, and anastomotic bleeding. Accordingly, many anesthesiologists have been seeking methods through which such laryngeal irritation can be attenuated, thus allowing for a smoother extubation. Furthermore, it has contributed to the aggravation of cough reflexes.

DETAILED DESCRIPTION:
Several strategies have been reported to facilitate smoother extubation, such as intravenous lidocaine, remifentanil, and dexmedetomidine. Dexmedetomidine is a potent, alpha-2-selective adrenoceptor agonist that causes sympatholytic, sedation and analgesia without respiratory compromise. The sedative properties of dexmedetomidine are largely due to effects on the locus ceruleus, producing a level of consciousness mimicking natural sleep Delivering dexmedetomidine intravenously to attenuate airway and circulatory reflexes during extubation has been extensively evaluated in clinical studies. Recent studies have also indicated that the intranasal application of dexmedetomidine is significantly useful and effective in the achievement of improved sedation and analgesia) and offers a safety profile similar to traditional sedatives ( ketamine and midazolam). Additionally, intratracheal local anesthetic instillation has been reported to be effective in preventing laryngeal reflexes. However, both the efficacy and safety profile of intratracheal dexmedetomidine applications are largely unknown and the technique has not been specifically investigated.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status classification I-II.
* Scheduled for lower abdominal surgeries e.g. congenital hernia repair and correction of penile hypospadias under general anesthesia (GA).

Exclusion Criteria:

* Younger than 1 year and older than 6 years of age,
* ASA score of III to IV.
* Parental refusal
* Allergy or contraindication to studied medication or anesthetic agents
* Patients with respiratory disease, heart disorders which might represent risk factors of potential complications of Dexmedetomidine such as bradycardia, hepatic or renal insufficiency.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
the coughing severity | intraoperative (during the recovery period from the time of awareness to 5 min after extubation)
  judged by the 4-point scale. 0 = no cough, 1= minimal (single) cough, 2 = moderate (≤5 ) cough and 3= severe (>5 ) cough.
  Grades 2 and 3 were bad.

SECONDARY OUTCOMES:
the Pediatric Objective Pain Scale | 24 hours postoperative
  monitor pain in children after surgery.• Minimum score: 0
  * Maximum score: 10
  * Maximum score if too young to complain of pain: 8
  * The higher the score the greater the degree of pain

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut governorate, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fan Q, Hu C, Ye M, Shen X. Dexmedetomidine for tracheal extubation in deeply anesthetized adult patients after otologic surgery: a comparison with remifentanil. BMC Anesthesiol. 2015 Jul 23;15:106. doi: 10.1186/s12871-015-0088-7. PMID 26202786
- [Background] Bhattacharjee DP, Saha S, Paul S, Roychowdhary S, Mondal S, Paul S. A comparative study of esmolol and dexmedetomidine on hemodynamic responses to carbon dioxide pneumoperitoneum during laparoscopic surgery. Anesth Essays Res. 2016 Sep-Dec;10(3):580-584. doi: 10.4103/0259-1162.183564. PMID 27746555
- [Background] Kim H, Min KT, Lee JR, Ha SH, Lee WK, Seo JH, Choi SH. Comparison of Dexmedetomidine and Remifentanil on Airway Reflex and Hemodynamic Changes during Recovery after Craniotomy. Yonsei Med J. 2016 Jul;57(4):980-6. doi: 10.3349/ymj.2016.57.4.980. PMID 27189295